CLINICAL TRIAL: NCT03087110
Title: Safety Study of Sibling Cord Blood Cell Infusion to Children With Cerebral Palsy
Brief Title: Stem Cells in Umbilical Blood Infusion for CP
Acronym: SCUBI-CP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other); Children's Health Queensland (Unknown); Monash Health (Other); Sydney Children's Hospitals Network (Other); Cerebral Palsy Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC/14/RCHM/38; RCH ID 34210; U1111-1179-9253 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2017-02-26; First posted 2017-03-22 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cord blood infusion (Experimental): Matched sibling donor cord blood cell infusion
  Interventions: Biological: Matched sibling donor cord blood cell infusion

INTERVENTIONS:
Biological: Matched sibling donor cord blood cell infusion — Single dose intravenous infusion of 12/12 HLA matched sibling donor cord blood cells (>1x10^7 cells/kg)

SUMMARY:
This study will investigate the safety of single dose intravenous infusion of cord blood cells which were cryopreserved after the birth of a brother or sister to a child with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common physical disability of childhood, affecting 2 per 1000 live births across the world. CP describes permanent non-progressive motor disorders arising from damage to the developing brain.

Preclinical studies of different types of stem cells in models of acute brain injury similar to CP have shown significant functional improvement. The variety of stem cells available in umbilical cord blood (UCB), an ethically uncomplicated source of stem cells, has led to a focus on UCB stem cell therapy as a quick-to-clinic option. Previous studies indicate that autologous or unrelated donor UCBC infusion is safe and feasible for children with CP, and may lead to improved motor functioning, but there is no information about the safety and effects of matched sibling cord blood. Therefore, this trial will study the safety of infusing matched sibling cord blood cells to children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of any type of CP
2. CP of any severity
3. A record of sibling CBU in storage at a TGA accredited private cord blood bank
4. Ability to travel to one of the trial centres
5. Ability to participate in assessments
6. Informed consent by parent/guardian

Exclusion Criteria:

1. presence of progressive neurological disease
2. known genetic disorder
3. known brain dysplasia
4. immune system disorder or immune deficiency syndrome
5. infectious disease markers showing up on virology screen
6. evidence of cord blood unit contamination, or fewer than 10^7 cells/kg body mass
7. ventilator support
8. ill health, or if the participant's medical condition does not allow safe travel
9. previous cell therapy
10. Botulinum toxin A within 3 months before or after infusion
11. surgery within 3 months before or after infusion
12. cannot obtain parent/guardian consent

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal clinical assessment and/or laboratory values | 12 months
  Safety

SECONDARY OUTCOMES:
Preliminary analysis of change in gross motor function | Baseline, 3 months
  Gross Motor Function Measure (GMFM-66)
Preliminary analysis of change in gross motor function | Baseline, 12 months
  Gross Motor Function Measure (GMFM-66)
Preliminary analysis of change in fine motor function | Baseline, 3 months
  Quality of Upper Extremity Skills Test (QUEST)
Preliminary analysis of change in fine motor function | Baseline, 12 months
  Quality of Upper Extremity Skills Test (QUEST)
Preliminary analysis of change in cognitive function | Baseline, 12 months
  Age appropriate cognitive testing: Bayley Scales of Infant and Toddler Development (BSID-III), Wechsler Preschool Primary Scale of Intelligence (WPPSI-IV), Wechsler Intelligence Scale for Children (WISC-V). Change from baseline will be compared using z-scores across measures.
Preliminary analysis of change in quality of life | Baseline, 3 months
  Cerebral Palsy Quality of Life (CP-QoL-CHILD)
Preliminary analysis of change in quality of life | Baseline,12 months
  Cerebral Palsy Quality of Life (CP-QoL-CHILD)
Digital PCR analysis of peripheral blood cellular DNA to determine the fraction of donor DNA in circulation | 3 months
  Chimerism study to detect the longevity of infused cells

CONTACTS AND LOCATIONS:
Overall Officials: Dinah Reddihough, MBChB, MD, Principal Investigator — Group leader
Locations (2):
- Australia (2):
  - Lady Cilento Children's Hospital, Brisbane, Queensland
  - The Royal Children's Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the SCUBI-CP trial will be available six months after publication of the primary outcome. The study protocol, analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute. Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the SCUBI-CP Trial Steering Committee must see and approve the analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgement and any additional costs involved must be covered. Should the Trial Steering Committee be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognised research institution which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary outcome
Access Criteria: 1) Data access agreement; 2) approval by Trial Steering Committee; 3) recognised research institutions.

REFERENCES:
- [Derived] Crompton K, Novak I, Fahey M, Badawi N, Lee KJ, Mechinaud-Heloury F, Edwards P, Colditz P, Soosay Raj T, Hough J, Wang X, Paget S, Hsiao KC, Anderson P, Reddihough D. Safety of sibling cord blood cell infusion for children with cerebral palsy. Cytotherapy. 2022 Sep;24(9):931-939. doi: 10.1016/j.jcyt.2022.01.003. Epub 2022 Feb 19. PMID 35193825
- [Derived] Crompton K, Novak I, Fahey M, Badawi N, Wallace E, Lee K, Mechinaud-Heloury F, Colditz PB, Elwood N, Edwards P, Reddihough D. Single group multisite safety trial of sibling cord blood cell infusion to children with cerebral palsy: study protocol and rationale. BMJ Open. 2020 Mar 8;10(3):e034974. doi: 10.1136/bmjopen-2019-034974. PMID 32152173

DOCUMENTS (1):
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT03087110/Prot_000.pdf